CLINICAL TRIAL: NCT03152214
Title: Physical Activity and Community Engagement (PACE) Among Returning Veterans
Acronym: PACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Team Red, White, and Blue (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-03-0109
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Reintegration
Keywords: Transition out of military

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Team RWB + Vigorous Intensity Aerobic Exercise (Experimental): Participants assigned to the integrated arm will be prescribed the following for the course of 8 weeks:
  * 1 session of exercise counseling
  * 3 weekly 25-minute sessions of vigorous intensity aerobic exercise
  * 1 weekly Team RWB event
  * 4 biweekly assessments
  Participants will also complete an online assessment at week 9 to provide follow-up data.
  Interventions: Other: Vigorous Intensity Aerobic Exercise and Community Engagement
- Team RWB (Active Comparator): Participants assigned to the Team RWB arm will be prescribed the following for the course of 8 weeks:
  * 1 weekly Team RWB event
  * 4 biweekly assessments
  Participants will also complete an online assessment at week 9 to provide follow-up data.
  Interventions: Other: Community Engagement
- Waitlist (No Intervention): Participants assigned to the waitlist arm will be prescribed the following for the course of 8 weeks:
  • 4 biweekly assessments
  Participants will also complete an online assessment at week 9 to provide follow-up data.

INTERVENTIONS:
Other: Vigorous Intensity Aerobic Exercise and Community Engagement — Each veteran will be provided with an Apple watch for the duration of the study. Research staff will use the resultant data to monitor the veteran's activity level. Veterans will be asked to complete three 25-minute sessions of vigorous intensity aerobic exercise per week (either running, cycling, rowing, or elliptical workouts). Data collected will include the number of minutes exercised and the heartrate level (77-85% maximum heart rate). Any exercise session of 25 minutes at > 76% of maximum heart rate will be characterized as 1 completed session of vigorous-intensity exercise. Veterans will enter the activity, minutes exercised, average heartrate, and perceived exertion into REDCap.
  Community engagement will involve attending at least one Team RWB event per week through the Austin or Killeen chapters. This could be a weekly running group, hike, or community service project-among other activities. Veterans will enter whether or not they attended a Team RWB event on REDCap.
  Arms: Team RWB + Vigorous Intensity Aerobic Exercise
Other: Community Engagement — Veterans in the study will receive a monthly calendar of Team RWB events upon assignment. Veterans will be able to participate in any Team RWB event located in Austin or Killeen. Veterans will be asked to attend at least one Team RWB event. This could be a weekly running group, hike, or community service project- among other activities. Veterans will enter whether or not they attended a Team RWB event on the REDCap exercise adherence surveys.
  Arms: Team RWB

SUMMARY:
Over 2 million soldiers have deployed during the Operation Enduring Freedom (OEF) and Operation Iraqi Freedom (OIF) conflicts. While the majority of veterans reintegrate successfully following deployment, a sizable minority return and face difficulties transitioning into civilian life. There is surprisingly little research on disseminable programs to facilitate reintegration, particularly outside of the formal VA healthcare system. The primary objective of this project is to develop and evaluate an integrated community- and exercise-based program that can be "prescribed" to augment existing transition assistance programs.

DETAILED DESCRIPTION:
Founded in 2010, Team Red White and Blue (RWB) is a non-profit organization that aims to enrich the lives of veterans by enhancing their connection to their community. Initial survey findings support the mission by showing that involvement in Team RWB (1) increases connectivity; (2) helps bridge the civilian/military divide; and (3) improves well-being and life satisfaction.

Numerous trials indicate that engaging in exercise programs can improve mood and reduce symptoms of depression and anxiety (for review see Penedo and Dahn, 2005). Accordingly, prescribing a structured exercise program has the potential to facilitate involvement in RWB and a reduction in reintegration difficulties. Compared to other levels of exercise intensity, vigorous-intensity exercise has been associated with increases in well-being (Cox, Thomas, Hinton, Donahue, 2006), reductions in anxiety and depression (Balchin, Linde, Blackhurst, Rauch, & Schönbächler, 2016; Cox, Thomas, Hinton, & Donahue, 2004; Katula, Blissmer, & McAuley, 1999) and improvements in quality of life (Ostman, Jewiss, & Smart, 2016). According to the American College of Sports Medicine (ACSM), high intensity exercise methods are the leading trend in the fitness industry (Thompson, 2013). Importantly, high intensity exercise programs have gained increasing popularity particularly within military units (Haddock, Poston, Heinrich, Jahnke, & Jitnarin, 2016).

This study aims to provide a pilot test of (1) the acceptability and effectiveness of RWB for veterans transitioning out of the military and (2) the effectiveness of a vigorous-intensity aerobic exercise prescription for enhancing the efficacy of RWB. To this end, the study will be a randomized controlled trial (RCT) that involves 75 veterans discharged from the US Army at Fort Hood who will be assigned to: 1) 8-weeks of vigorous-intensity aerobic exercise in addition to participation in a community-based program (Team RWB) or (2) 8-weeks of participation in Team RWB alone or (3) 8-weeks on a waitlist.

ELIGIBILITY:
Inclusion Criteria:

* OEF/OIF/OND veteran
* Discharged from the US Army within/up to 12 months ago
* Endorse at least moderate difficulty with reintegration (a total score of at least 1.5 on the M2C-Q and a score of 2 on item #14)
* Use or have access to an Apple iPhone
* Has participated in less than 75 minutes of vigorous-intensity exercise per week over the last two weeks
* Understanding and willingness to comply to a 9-week study protocol

Exclusion Criteria:

* Condition or injury which would prevent exercise*
* Insufficient command of the English language

Each veteran will complete the PAR-Q as part of the screening procedure in order to check for any condition/injury which would render exercise harmful. Each veteran will also have undergone a routine physical with medical staff prior to discharge from the U.S. Army. Thus, the veteran should have knowledge of a condition or injury which could be problematic. If such a risk is present, the veteran will be excluded from the study. Veterans will be excluded if a doctor has said that they have a heart condition and should not do physical activity or if they know of any other reason why they should not engage in physical activity. Veterans who are unsure if they are able to engage in physical activity will have to have signed approval from a physical.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Level of Reintegration Difficulties | 9 weeks
  The Military to Civilian Questionnaire (M2C-Q) is a 16-item self-report measure of post deployment community reintegration difficulty. The M2C-Q assesses a number of theoretically related domains (e.g., overall mental health, probably PTSD, separate rating of difficulty readjusting to civilian life; Sayer et al., 2011).

SECONDARY OUTCOMES:
Acceptability of the Intervention | 9 weeks
  This will be assessed by looking at adherence to exercise or Team RWB events. The investigators will also include a measure to assess veterans' perceptions of the exercise program and of Team RWB in terms of likelihood of future engagement, program likeability, and perceived benefits of the intervention.
Meaning in life | 9 weeks
  The Meaning in Life Questionnaire (MLQ) is a 10-item measure designed to measure two dimensions of meaning in life: 1) presence of meaning (how much participants feel that their lives have meaning) and 2) search for meaning (how much participants strive to find meaning in their lives).
Depressive Symptoms | 9 weeks
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item measure designed to screen for and monitor the severity of depressive symptoms.
Life Satisfaction | 9 weeks
  The Satisfaction with Life Scale (SWLS) is a 5-item instrument designed to measure global cognitive judgments of satisfaction with one's life (Diener, Emmons, Larsen, & Griffin, 1985).
Life Enrichment | 9 weeks
  The Team RWB Enriched Life Scale (ELS) is a 48-item instrument designed to measure an "enriched" life defined as positive health, genuine relationships, and sense of individual and shared purpose.

CONTACTS AND LOCATIONS:
Overall Officials: Scarlett O Baird, M.A., Principal Investigator — University of Texas at Austin; Jasper A Smits, Ph.D., Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States